CLINICAL TRIAL: NCT01114204
Title: A Phase III, Randomized, Open-label, Active-Controlled, Trial Comparing Ferumoxytol With Iron Sucrose for the Treatment of Iron Deficiency Anemia
Brief Title: A Trial Comparing Ferumoxytol With Iron Sucrose for the Treatment of Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-FER-IDA-302
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; Feraheme; ferumoxytol; iron sucrose; Venofer; IDA
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferumoxytol (Experimental): Participants received a total of 2 doses of IV ferumoxytol 510 milligrams (mg) (17 milliliters [mL]). The first IV 510 mg dose was administered on Day 1 (Baseline) and second dose 2 to 8 (5±3) days after the first dose, for a total cumulative dose of 1.02 grams (g).
  Interventions: Drug: Ferumoxytol
- Iron Sucrose (Active Comparator): Participants received an IV injection or infusion of iron sucrose 200 mg (10 mL) on Day 1 (Baseline) and on 4 other non-consecutive days over a 14-day period, for a total cumulative dose of 1.0 g. Participants receiving their first ever exposure to IV iron sucrose, received a test dose on Day 1 prior to receiving the remainder of the first dose, as prescribed in the package insert for some countries.
  Interventions: Drug: Iron Sucrose

INTERVENTIONS:
Drug: Ferumoxytol — IV Ferumoxytol
  Other Names: Feraheme
  Arms: Ferumoxytol
Drug: Iron Sucrose — IV Iron Sucrose
  Other Names: Venofer
  Arms: Iron Sucrose

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of intravenous (IV) ferumoxytol compared to IV iron sucrose for the treatment of iron deficiency anemia (IDA).

ELIGIBILITY:
Key Inclusion Criteria include:

1. Males and females ≥18 years of age
2. Participants with IDA defined as having:

   1. Hemoglobin <10.0 g/deciliter (dL)
   2. Transferrin saturation (TSAT) <20%
3. Participants who have a history of unsatisfactory oral iron therapy or in whom oral iron cannot be used
4. Female participants of childbearing potential who are sexually active must be on an effective method of birth control for at least 1 month prior to screening and agree to remain on birth control until completion of participation in the study

Key Exclusion Criteria include:

1. History of allergy to IV iron
2. Allergy to two or more classes of drugs
3. Participants on dialysis or with an estimated glomerular filtration rate <30 mL/minute(min)/1.73 square meter (m^2)
4. Female participants who are pregnant, intend to become pregnant, are breastfeeding, within 2 weeks postpartum, or have a positive serum/urine pregnancy test
5. Hemoglobin ≤7.0 g/dL
6. Serum ferritin >600 nanogram/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2010-08-10 (Actual); Primary Completion 2011-11-09 (Actual); Study Completion 2012-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- Australia (7):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ballarat
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Five Dock
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gosford
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingswood
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville
- For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Tronche, France
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siegen
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilhelmshaven
- Hungary (8):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Békéscsaba
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Komárom
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miskolc
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szekszárd
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vác
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
- Latvia (4):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daugavpils
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riga
  - For additional this triinformation regarding investigative sites for al, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riga
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ventspils
- Lithuania (4):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipėda
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Šiauliai
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sopot
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zgierz
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Łęczyca
- Romania (6):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suceava
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- South Africa (4):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roodepoort
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheonan
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manresa
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Cruz de Tenerife
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Ukraine (9):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherkasy
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chernivtsi
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivano-Frankivsk
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Simferopol
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaporizhzhya
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Background] Strauss WE, Dahl NV, Li Z, Lau G, Allen LF. Ferumoxytol versus iron sucrose treatment: a post-hoc analysis of randomized controlled trials in patients with varying renal function and iron deficiency anemia. BMC Hematol. 2016 Jul 26;16:20. doi: 10.1186/s12878-016-0060-x. eCollection 2016. PMID 27462400
- [Background] Hetzel D, Strauss W, Bernard K, Li Z, Urboniene A, Allen LF. A Phase III, randomized, open-label trial of ferumoxytol compared with iron sucrose for the treatment of iron deficiency anemia in patients with a history of unsatisfactory oral iron therapy. Am J Hematol. 2014 Jun;89(6):646-50. doi: 10.1002/ajh.23712. PMID 24639149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to enrollment for adult participants with iron deficiency anemia (IDA), defined as hemoglobin <10.0 grams (g)/deciliter (dL) and transferrin saturation (TSAT) <20%, and a history of unsatisfactory oral iron therapy or in whom oral iron could not be used.
Groups:
- Ferumoxytol: Participants received a total of 2 doses of intravenous (IV) ferumoxytol 510 milligrams (mg) (17 milliliters [mL]). The first IV 510 mg dose was administered on Day 1 (Baseline) and second dose 2 to 8 (5±3) days after the first dose, for a total cumulative dose of 1.02 g.
Period: Overall Study
Arm/Group | Ferumoxytol | Iron Sucrose
Started | 406 | 199
Received at Least 1 Dose of Study Drug | 406 | 199
Completed (Completed is defined as had study drug and Week 5 visit.) | 385 | 191
Not Completed | 21 | 8
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Death | 1 | 0
Not completed — Other-Personal reasons | 2 | 0
Not completed — Other-Medical monitor request | 1 | 0
Not completed — Other-Participant request | 2 | 0
Not completed — Other-Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: Any randomized participant who had any exposure to study drug (ferumoxytol or iron sucrose) and was based upon randomized treatment assignment.
Groups:
- Ferumoxytol: Participants received a total of 2 doses of IV ferumoxytol 510 mg (17 mL). The first IV 510 mg dose was administered on Day 1 (Baseline) and second dose 2 to 8 (5±3) days after the first dose, for a total cumulative dose of 1.02 g.
- Iron Sucrose: Participants received an IV injection or infusion of iron sucrose 200 mg (10 mL) on Day 1 (Baseline) and on 4 other non-consecutive days over a 14-day period for a total cumulative dose of 1.0 g. Participants receiving their first ever exposure to IV iron sucrose, received a test dose on Day 1 prior to receiving the remainder of the first dose, as prescribed in the package insert for some countries.
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol | Iron Sucrose | Total
Number analyzed (Participants) | 406 | 199 | 605
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (14.89) | 48.9 (14.66) | 48.2 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 342 | 160 | 502
  Male | 64 | 39 | 103

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieved A ≥2.0 g/dL Increase In Hemoglobin At Any Time From Baseline To Week 5
Description: Participants who achieved a ≥2.0 g/dL increase in hemoglobin at any time from Baseline up to Week 5 are presented. Increase in hemoglobin at any time from Baseline up to Week 5 was calculated for each participant based on:
  Hemoglobin Change = Hemoglobin (Week X) - Hemoglobin (Baseline), where Week X was any post-Baseline visit up to and including Week 5.
  Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. Participants with no post-Baseline hemoglobin values were classified as not achieving a ≥2.0 g/dL increase.
  Statistical analysis was performed for data up to Week 5 only.
Time Frame: Baseline (Day 1) through Week 5
Population: ITT Population: Any randomized participant who had any exposure to study drug (ferumoxytol or iron sucrose) and was based upon randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 406 | 199
Participants
  Up to Week 3 | 291 | 117
  Up to Week 4 | 327 | 145
  Up to Week 5 | 341 | 162
Statistical Analysis 1: Comparison: Ferumoxytol vs Iron Sucrose; Participants who achieved a ≥2.0 g/dL increase in hemoglobin from Baseline up to Week 5 were analyzed. Statistical comparison was performed for data up to Week 5 only. Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information; Test type: Non-Inferiority — The 95% confidence interval (CI) was calculated using the large sample assumption. The pre-defined non-inferiority margin for testing the difference between treatment groups was -15%; p = 0.2833, Cochran-Mantel-Haenszel; The p-value is the result of the Cochran-Mantel-Haenszel test, adjusted for Baseline hemoglobin level and underlying condition; Treatment Difference = 2.58, 95% CI 2-sided [-3.89 to 9.06] — The treatment difference (ferumoxytol - iron sucrose) was expressed as a percentage

2. Secondary Outcome: Mean Change In Hemoglobin From Baseline To Week 5
Description: Mean change in hemoglobin from Baseline to Week 5 was calculated for each participant as: Hemoglobin Change = Hemoglobin (Week 5) - Hemoglobin (Baseline).
  Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. If the Week 5 hemoglobin value was missing, the change from Baseline was imputed to be zero.
Time Frame: Baseline (Day 1), Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 406 | 199
g/dL | 2.9 (1.62) | 2.7 (1.30)

3. Secondary Outcome: Participants Achieving A Hemoglobin Level ≥12.0 g/dL At Any Time From Baseline To Week 5
Description: Participants who achieved a ≥12.0 g/dL hemoglobin level at any time from Baseline up to Week 5 are presented. Increase in hemoglobin at any time from Baseline up to Week 5 was calculated for each participant based on:
  Hemoglobin Change = Hemoglobin (Week X) - Hemoglobin (Baseline), where Week X was any post-Baseline visit up to and including Week 5. Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. Participants without any post-Baseline hemoglobin values were treated as non-responders.
Time Frame: Baseline (Day 1) through Week 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 406 | 199
Participants
  Up to Week 3 | 123 | 33
  Up to Week 4 | 210 | 67
  Up to Week 5 | 271 | 96

4. Secondary Outcome: Mean Change In TSAT From Baseline To Week 5
Description: Mean change in TSAT from Baseline to Week 5 was calculated for each participant as: TSAT Change = TSAT (Week 5) - TSAT (Baseline).
  Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. If the Week 5 TSAT value was missing, the change from Baseline was imputed to be zero.
Time Frame: Baseline (Day 1), Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 406 | 199
percentage of saturation | 15.7 (16.80) | 11.9 (14.41)

5. Secondary Outcome: Mean Change In Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score From Baseline To Week 5
Description: The FACIT-Fatigue questionnaire is a 13 item questionnaire designed and validated to specifically assess the presence and impact of treatment on fatigue and related symptoms, such as tiredness, on health-related quality of life in anemic participants with cancer. The questionnaire has 13 items, each measured on a 4-point Likert scale. Scoring ranges from 0 (the most fatigued) to 52 (the least fatigued) points, with higher scores representing better functioning or less fatigue.
  Mean change in FACIT-Fatigue Score from Baseline to Week 5 was calculated for each participant as:
  FACIT-Fatigue Score Change = FACIT-Fatigue Score (Week 5) - FACIT-Fatigue Score (Baseline).
  Baseline was defined as the Day 1 value (prior to first dose of study drug).The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. If the Week 5 FACIT-Fatigue Score value was missing, the change from Baseline was imputed to be zero.
Time Frame: Baseline (Day 1), Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 399 | 198
units on a scale | 13.1 (11.78) | 12.4 (11.22)

6. Secondary Outcome: Time To Hemoglobin Increase Of ≥2.0 g/dL Or Hemoglobin Value Of ≥12.0 g/dL From Baseline
Description: The time to hemoglobin increase of ≥2.0 g/dL or hemoglobin value of ≥12.0 g/dL was defined as the days from Baseline (Day 1) to the first time the participant had an increase in hemoglobin of ≥2.0 g/dL or hemoglobin value of ≥12.0 g/dL, and was calculated using a Kaplan-Meier curve. Participants who did not have a hemoglobin increase of ≥2.0 g/dL or to a hemoglobin level ≥12.0 g/dL were censored at their last visit day. Participants without any post-Baseline study visits were not included.
Time Frame: From Baseline (Day 1) up to Week 5
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 406 | 199
days | 23.1 [15.0 to 24.0] | 25.2 [21.0 to 30.0]

ADVERSE EVENTS:
Arm/Group | Ferumoxytol | Iron Sucrose
Serious Adverse Events (participants affected / at risk) | 17/406 | 5/199
Other Adverse Events (participants affected / at risk) | 95/406 | 69/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ferumoxytol (N=406) | Iron Sucrose (N=199)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bartholin's abscess (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/342 | 0/160
Dysuria (Renal and urinary disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 2/342 | 0/160
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ferumoxytol (N=406) | Iron Sucrose (N=199)
Nausea (Gastrointestinal disorders) | 11 | 7
Dry mouth (Gastrointestinal disorders) | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 3 | 4
Chest discomfort (General disorders) | 9 | 2
Pyrexia (General disorders) | 2 | 6
Chills (General disorders) | 0 | 4
Urinary tract infection (Infections and infestations) | 2 | 3
Cystitis (Infections and infestations) | 1 | 3
Alanine aminotransferase increased (Investigations) | 4 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 3
White blood cell count decreased (Investigations) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Headache (Nervous system disorders) | 19 | 11
Dizziness (Nervous system disorders) | 9 | 3
Dysgeusia (Nervous system disorders) | 9 | 13
Dysmenorrhoea (Reproductive system and breast disorders) | 3/342 | 3/160
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Hypertension (Vascular disorders) | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 4 | 2
Fatigue (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 3 | 2
Feeling hot (General disorders) | 2 | 2
Injection site pain (General disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 3 | 2
Drug hypersensitivity (Immune system disorders) | 2 | 2
Influenza (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Lymphocyte count decreased (Investigations) | 4 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 2
Blood urea decreased (Investigations) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Somnolence (Nervous system disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data have been received by Sponsor, the Site, and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.